CLINICAL TRIAL: NCT00375544
Title: A Phase I Single Center Open Label Study to Evaluate the Safety and Efficacy of a Low Level Light Device in Patients With Knee Osteoarthritis
Brief Title: Study to Evaluate the Safety and Efficacy of a Low Level Light Device in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Sciences LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C00011
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Laser Therapy, Low-Level; Osteoarthritis; Phototherapy; Osteoarthritis, knee; Light-emitting diode
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Low-Level Light Therapy

INTERVENTIONS:
Device: Low level light therapy

SUMMARY:
This Phase I study is being conducted to examine the efficacy of the Light Sciences LLC (LSLLC) phototherapy device for home (self) treatment of knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This Phase I study is being conducted to examine the efficacy of the Light Sciences LLC (LSLLC) phototherapy device for home (self) - treatment of knee osteoarthritis (OA). Clinical efficacy will be assessed by evaluating the level of reported pain, including the use of analgesics, various measures of functional improvement, and clinical symptomology during a three week period of daily treatments. Durability of the clinical response for twelve weeks following therapy will also be examined. In addition, device safety will be assessed. As this is an early stage-prototype device, subject input regarding the usability of the device will be sought.

Subjects will be required to achieve three weeks of wash-out from all OA therapies prior to the start of phototherapy. Acetaminophen will be allowed during this time. During the three week active treatment and twelve week follow-up periods, subjects will be required to refrain from acetaminophen as well as OA therapies. However, subjects will be encouraged to speak with the investigator should any symptoms become difficult to manage. In addition to clinical assessments, subjects will be required to keep a daily diary.

The clinical objectives of the study will be met if at least five of ten subjects report decreased pain scores and improvement on an osteoarthritis index. While minimum or no safety issues are expected, the occurrence of skin changes to the area exposed to the device will be carefully monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* At least age 40 years
* Community ambulator without orthoses
* Knee circumference in range of 35.5 - 43 cm. (14-17 inches)
* Moderate OA according to clinician judgment, and/or Radiographic evidence of knee OA of Kellgren-Lawrence Grade II or III in one or both knees.
* Exercise induced pain, or for subjects who do not exercise, pain resulting from the activities of daily living, of at least 3 months duration
* Knee pain of greater than 1 on VAS within the last 24 hours before evaluation.
* Fitzpatrick type I, II, or III skin. (very light to darker Caucasian/light Asian.) (Selection avoids excessive light absorption in epidermis)
* Understands and agrees to comply with all study procedures including the daily treatments and follow-up visits
* Able to understand and is voluntarily willing to sign an informed consent form for this study

Exclusion Criteria:

* Pregnant or nursing, or with the ability to become pregnant and not using an accepted form of birth control
* Other causes of knee-related pain (e.g. hip OA, arterial insufficiency, etc) have been ruled out by physical examinations
* Fitzpatrick type IV, V, or VI skin. (Mediterranean/Asian/Hispanic to dark-skinned black)
* Any active Cancer
* History of melanoma to the limb that is being evaluated in this study
* Uncontrolled diabetes mellitus
* Untreated hypertension
* Skin conditions that would interfere with device use/placement
* Psychotic disorder(s), dementia, mental retardation, or other organic mental disorders (subjects who are not mentally and physically able to personally consent for participation in this study are not eligible)
* Any other (including acute) condition, which in the opinion of the investigator, is likely to cause non-compliance or significantly impact treatment outcomes.
* Subject has received intra- or peri- articular steroid, or other, injection therapy within 6 months prior to enrollment in this study.
* Enrolled in any other clinical trial within the last 6 weeks or enrollment in another clinical trial during participation in this trial.

Subjects who cannot be expected to be able to comply with the following restrictions during the course of their participation in the study, including during the washout period:

* Prescription NSAID use prohibited
* Use of photosensitizing drugs prohibited
* Physiotherapy prohibited for treatment to the limb(s) that is being evaluated in this study.
* Glucosamine use prohibited

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Decreased pain scores on the visual analog scale (VAS)
Improved Western Ontario and McMaster Universities Osteoarthritis index (WOMAC) scores

SECONDARY OUTCOMES:
Reduced use of over the counter (OTC) analgesics post therapy
Improved functionality as determined by measurable increases in knee range of motion (ROM)
Increased exercise ability
No, or decreased knee effusion
Subject satisfaction
Durability of the Clinical Response

CONTACTS AND LOCATIONS:
Overall Officials: James C Chen, M.D., Study Director — Light Sciences LLC
Locations (1):
- Richard Neiman, M.D., Kirkland, Washington, United States